CLINICAL TRIAL: NCT04846023
Title: Pediatric Delirium Screening in the PICU Via EEG
Acronym: PEDEEGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Laurence Ducharme-Crevier, Pediatric intensivist, Principal Investigator, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSJ-2021-xxx
Record Dates: First submitted 2021-04-01; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: Single center prospective interventional study of children admitted to a PICU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amplitude EEG (aEEG) via VEEGix (Experimental): Amplitude-Integrated EEG can be achieved with a limited number of frontal electrodes.
  Interventions: Device: aEEG via vEEGix

INTERVENTIONS:
Device: aEEG via vEEGix — Amplitude-Integrated EEG can be achieved with a limited number of frontal electrodes. There is a new aEEG technology available: VEEGix, developed by NeuroServo Inc. It is a miniaturized aEEG, non-intrusive, portable and resistant to patient's movements. Its main advantage is its simplicity of use as a single adhesive strip including all electrodes is fixed to the patient's forehead and is connected to the VEEGix device

SUMMARY:
Delirium in the pediatric intensive care unit (PICU) is a serious problem that has recently attracted much attention. This study will evaluate the use of electroencephalogram (EEG) for delirium screening in the PICU.

DETAILED DESCRIPTION:
Primary objective: In a prospective cohort of children hospitalized in a PICU, EEG features associated with pediatric delirium (via VEEGix) will be identified and the diagnostic value to accurately detect delirium of these features will be calculated.

Secondary objective: To investigate the accuracy and rapidity of delirium diagnosis with the VEEGix.

ELIGIBILITY:
Inclusion Criteria:

Eligible for inclusion children 1) <18 years; and 2) admitted to the PICU at the Centre Hospitalier Universitaire Ste-Justine (CHUSJ). To select patients at high risk for delirium, one of the following inclusion criteria will be needed: 3) mechanically ventilated patients; or 4) non-invasively ventilated patients (BiPap, Cpap or high flow nasal cannula); or 5) patients receiving opioids; or 6) patients receiving benzodiazepines.

Exclusion Criteria:

Children 1) suspected of being brain death at the time of PICU entry (Glasgow Coma Scale (GCS) 3 and loss of all brain stem reflexes); 2) with significant clinical developmental delay (based on clinical assessment and/or parental report of developmental problems that affected the child's behavior or ability to communicate; Pediatric Cerebral Performance Category ≥4); 3) planned discharge from the PICU the same or next day.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
In a prospective cohort of children hospitalized in a PICU, the EEG features associated with pediatric delirium (via VEEGix) willl be identified. | 1 year recruitment
  Variables will include 1) predominant background frequencies: delta 0-3.9 Hz, theta 4-7.9 Hz, alpha 8-11.9 Hz and beta 12-30 Hz and power spectrum (ratio of each frequency/total 0-30Hz), 2) EEG: symmetry (symmetric, mild asymmetry, marked asymmetry) and prevalence (continuous, nearly continuous (1-9% of suppression or attenuation), discontinuous (10-49% of suppression or attenuation), burst suppression or burst-attenuation (50-99% of suppression or attenuation), suppression (>99% of suppression or attenuation) as measured by percentage per hour of recording)(19). As power across all frequency bands decreases significantly with age, children will be divided 0 to 6 months, 6 months to 3 years and 3-18 years old.

SECONDARY OUTCOMES:
To investigate the accuracy and rapidity of delirium diagnosis with the VEEGix. | 1 year recruitment
  The diagnosis of delirium by the vEEGix will be defined as presence of EEG characteristics of delirium (identified in objective 1). Diagnosis of delirium by the vEEGix will be compared to the diagnosis of delirium by the medical team (confirmed by a adjudicating committee). Timing of delirium diagnosis will be compared: diagnosis by the medical team (defined as the first CAPD scores equal or greater than 9) versus diagnosis by the vEEGix (the beginning of the delirium episode will be defined as the appearance of these EEG characteristics).

IPD SHARING:
Plan to Share IPD: No